CLINICAL TRIAL: NCT05799560
Title: Determination of the Effect of Therapeutic Touch and Reiki Application on Anxiety and Stress Levels in Female Academicians
Brief Title: The Effect of Therapeutic Touch and Reiki Application on Anxiety and Stress Levels in Female Academicians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Emine Yıldırım, Assistant Professor, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: p3s5qeux
Record Dates: First submitted 2023-01-10; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Stress; Anxiety
Keywords: academics; therapeutic touch; reiki
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention
- intervention (Experimental): Reiki touch and terapotic touch will be done
  Interventions: Other: THERAPEUTIC TOUCH; Other: REİKİ

INTERVENTIONS:
Other: THERAPEUTIC TOUCH — Therapeutic touch will be done. It will be applied twice a week for two weeks, each application for 20 minutes.
  Arms: intervention
Other: REİKİ — It will be applied twice a week for two weeks, each application for 20 minutes.
  Arms: intervention

SUMMARY:
Stress and anxiety form an integral part of organizational life in universities. Studies reveal that the stress experienced by academicians has increased dramatically in recent years. Stress affects employee performance. In order to reduce the stress level of female academicians, methods such as non-pharmacological treatment, massage that can be applied to support scientific medicine, acupressure, hot and cold application, therapeutic touch should be used. The non-pharmacological methods that investigators will look at in our research are therapeutic touch and reiki. The improvement of the balance in the body and the reduction of negative effects such as pain, stress and anxiety with non-pharmacological touch methods are explained by Gate Control and Endorphin theories. The universe of the research will be female academicians working at Osmaniye Korkut Ata University. participants will be determined by the block randomization method. Data; It will be collected using the Introductory Information Form, Depression, Anxiety and Stress Level Assessment Form. TT and Reiki application will have positive contributions as it is a non-pharmacological method, easy to apply and low cost. When the studies were examined, no other study was found in the same application as our study.

Therefore, in this study, it was aimed to evaluate the effect of therapeutic touch and reiki practice on anxiety and stress levels in female academicians.

ELIGIBILITY:
Inclusion Criteria:

* Academicians who do not have any communication problems
* Do not have psychological problems

Exclusion Criteria:

* Those who do not want to participate in the research

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-20 (Estimated)

PRIMARY OUTCOMES:
Depression Anxiety Stress Scale | 4 week
  The Dass-21 scale consists of 21 items that examine depression, anxiety and stress under three headings.
  This scale is a 4-point Likert-type scale and consists of 7 questions each measuring "depression, stress and anxiety dimensions".
  Subjects are asked to mark four different score types (0, 1, 2, and 3) opposite to each sentence according to the severity and frequency of their feelings, how they have felt in the last few weeks.
  If the given sentence does not fit the person at all, it is required to mark 0, if it is a satellite to some extent, 1 if it is a satellite to some extent, 2 if it is a satellite to a significant degree, and 3 if it is exactly a satellite.
  Then, the scores for each scale are summed and depression, anxiety and stress scores are found.
  Getting 5 points or more from depression sub-dimension, 4 points or more from anxiety, 8 points or more from stress indicates that the individual has a related problem.